CLINICAL TRIAL: NCT04686617
Title: The Effect of Twelve Weeks of Mechanical Vibration on Root Resorption: A Micro-Ct Study
Brief Title: Effect of Mechanical Vibration on Root Resorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Hakan Yılmaz, Assistant Professor, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 13112012
Record Dates: First submitted 2020-12-17; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Vibration; Exposure

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No-force group (No Intervention): The right and left side first premolar teeth were randomly assigned (split-mouth design) so that mechanical vibration was applied in the buccal direction on one side and the other side was used as the premolar tooth control group. Oral B HummingBird device (Procter&Gamble, USA) with a modified tip was used for the application of vibration. The tip was positioned mid-buccally of teeth to perform buccally directed vibration. HummingBird is prescribed maximum period 0.00885s corresponding to 6800RPM or 113Hz of the motor. The vibration procedure was applied for 10mins/day during the period of 12 weeks. At the end of the 12th week, the first stage was completed and the first premolar teeth were extracted.
- Force Group (Active Comparator): The right and left side first premolar teeth were randomly assigned (split-mouth design) so that mechanical vibration was applied in the buccal direction to one side and the other side was used as the premolar tooth control group. As in no-force group, same device procedure was used for the application of vibration. Self-ligating Speed (Strite Industries, Cambridge, Ontario, Canada) tubes and brackets with 0.022×0.026 inch slots were bonded to the buccal surfaces of the right and left first molar teeth and first premolar teeth.150g of buccally directed forces, producing by a 0.017×0.025-in beta-titanium-molybdenum alloy (3M Unitek, Monrovia, Calif) cantilever spring, were applied to premolar teeth on both side.The force magnitude was measured with a strain gauge (Dentaurum). At the end of the 12th week, the first stage was completed and the first premolar teeth were extracted.
  Interventions: Diagnostic Test: Mechanical Vibration

INTERVENTIONS:
Diagnostic Test: Mechanical Vibration — Oral B HummingBird device (Procter&Gamble, USA) with a modified tip was used for the application of vibration. The tip was positioned mid-buccally of teeth to perform buccally directed vibration. HummingBird is prescribed maximum period 0.00885s corresponding to 6800RPM or 113Hz of the motor. The vibration procedure was applied for 10mins/day during the period of 12 weeks.
  Arms: Force Group

SUMMARY:
The aim of this study was to investigate the effect of mechanical vibration on root resorption with or without the application of orthodontic force.

Twenty patients who required maxillary premolar extractions as part of their orthodontic treatment were randomly separated into two groups of 10: no-force group and force group. Using a split-mouth procedure, each patient's maxillary first premolar teeth were randomly assigned as either vibration or control side in both groups. Buccally directed vibration of 113 Hz, using an Oral-B HummingBird device with a modified tip, was applied to the maxillary first premolar for 10 mins/day during 12 weeks. After the force application period, the maxillary first premolars were extracted and scanned with micro-computed tomography. Fiji(ImageJ) which made slice-by-slice quantitative volumetric measurements was used for resorption crater calculation. Total crater volumes was compared with Wilcoxon and Mann-Whitney U tests.

DETAILED DESCRIPTION:
The sample included 40 maxillary first premolars from 20 orthodontic patients (7 boys and 13 girls; range: 15.08-18.58 years; mean: 16.77 years) who required bilateral maxillary first premolar extractions as part of their orthodontic treatment. They were recruited according to strict selection criteria as described previously.These included need for bilateral maxillary first premolar extractions (necessitating moderate anchorage) and fixed appliance treatment; permanent dentition; completion of apexification; similar minimal crowding on each side of the maxillary arch; no previous orthodontic or orthopedic treatment; no unilateral or bilateral posterior crossbites; no craniofacial anomaly; no history of trauma, bruxism, or parafunction; no past or present signs and symptoms of periodontal disease; no significant medical history that would affect the development or structure of the teeth and jaws and any subsequent tooth movement; and no history of asthma. The sample size was calculated by using Piface 1.72, and guaranteed 82.56% power. This number was reached by considering the standard deviation of 0.46mm3 in our previous similar study. True difference of means was estimated at 0.2mm3, and type I error(α) was accepted as the standard value .05.

Ethics approval was obtained from the Ethics Committee of Bulent Ecevit University (2012/23). All subjects and their guardians consented to participate in this study after receiving verbal and written explanations.

Impressions were taken with alginate of the maxillary jaw only to construct the appliance. The study model was obtained by pouring hard plaster. On this model, the transpalatal arch was formed by bending a 0.09 mm steel wire between the maxillary right and left first molar teeth. To prevent potential contact of the teeth during buccal movement to the transpalatal arch, occlusion rising acrylic plates were added. The acrylic plates were of mean 2mm thickness to only include occlusion of the first molar teeth. After fitting the transpalatal arches in the mouth, light-cured glass ionomer cement (TransbondTM Plus, 3M Unitek, Monrovia, USA) was applied to the maxillary first molar teeth of all the patients. After these procedures, the patients were randomly separated into 2 equal groups. Randomization was made using the Excel program (Microsoft, Redmond, WA, USA), and allocation was hidden in consecutively numbered, closed envelopes. Blinding was used for treatment and outcome assessments.

No-force group: The right and left side first premolar teeth were randomly assigned (split-mouth design) so that mechanical vibration was applied in the buccal direction on one side and the other side was used as the premolar tooth control group. Oral B Hummingbird device (Procter&Gamble, USA) with a modified tip was used for the application of vibration. The tip was positioned mid-buccally of teeth to perform buccally directed vibration. HummingBird is prescribed maximum period 0.00885s corresponding to 6800RPM or 113Hz of the motor. The vibration procedure was applied for 10mins/day during the period of 12 weeks. At the end of the 12th week, the first stage was completed and the first premolar teeth were extracted.

Force group: The right and left side first premolar teeth were randomly assigned (split-mouth design) so that mechanical vibration was applied in the buccal direction to one side and the other side was used as the premolar tooth control group. As in no-force group, same device procedure was used for the application of vibration. Self-ligating Speed (Strite Industries, Cambridge, Ontario, Canada) tubes and brackets with 0.022×0.026 inch slots were bonded to the buccal surfaces of the right and left first molar teeth and first premolar teeth.150g of buccally directed forces, producing by a 0.017×0.025-in beta-titanium-molybdenum alloy (3M Unitek, Monrovia, Calif) cantilever spring, were applied to premolar teeth on both side. The force magnitude was measured with a strain gauge (Dentaurum). At the end of the 12th week, the first stage was completed and the first premolar teeth were extracted.

The premolar teeth were extracted under local anesthesia by the same dental practitioner in all cases. To remove blood and tissue remnants from the teeth after extraction, they were washed with non-pressurized isotonic solution without touching the root surfaces, then each tooth was placed in a 5 ml sterile tube containing 10% formalin solution (Sarstedt Ag & Co., Nümbrecht, Germany). After 2 weeks the formalin solution was changed and no other procedure was applied until examination of the roots.

Scanning of the root surfaces was applied using the SkyScan-1172 x-ray micro-tomography device (SkyScan, Aartselaar, Belgium). To calculate the volume of the resorption craters isolated on the axial slices, open-source Fiji (ImageJ) software was used. Using the convex hull module in the software, a line was drawn joining the edges of the resorption craters and the area below the line was calculated as the volume (Figure 4). Volumetric changes in the craters on the root surfaces were evaluated both locally and totally.

The data were statistically analyzed using SPSS version 24.0(IBM Corp., Armonk, NY, USA). The Shapiro-Wilk test was used to test for normal distribution. Wilcoxon test was applied to the within-group comparisons of the resorption volumes formed at different levels(cervical, mid, apical) on different surfaces of the root(buccal, palatal, mesial, and distal). The Mann-Whitney U-test was used in comparisons between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Need for bilateral maxillary first premolar extractions (necessitating moderate anchorage) and fixed appliance treatment
* Permanent dentition
* Completion of apexification
* Similar minimal crowding on each side of the maxillary arch

Exclusion Criteria:

* Previous orthodontic or orthopedic treatment
* Unilateral or bilateral posterior crossbites
* Craniofacial anomaly
* History of trauma, bruxism, or parafunction
* Past or present signs and symptoms of periodontal disease
* Significant medical history that would affect the development or structure of the teeth and jaws and any subsequent tooth movement
* History of asthma

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Orthodontically induced inflammatory root resorption (OIIRR) | 12 weeks
  Orthodontically induced inflammatory root resorption (OIIRR) or, as it is better known, root resorption, is an unavoidable pathologic consequence of orthodontic tooth movement. It is a certain adverse effect of an otherwise predictable force application.

IPD SHARING:
Plan to Share IPD: Undecided
We can share when it's really needed.

REFERENCES:
- [Background] DiBiase AT, Woodhouse NR, Papageorgiou SN, Johnson N, Slipper C, Grant J, Alsaleh M, Khaja Y, Cobourne MT. Effects of supplemental vibrational force on space closure, treatment duration, and occlusal outcome: A multicenter randomized clinical trial. Am J Orthod Dentofacial Orthop. 2018 Apr;153(4):469-480.e4. doi: 10.1016/j.ajodo.2017.10.021. PMID 29602338
- [Background] Liao Z, Elekdag-Turk S, Turk T, Grove J, Dalci O, Chen J, Zheng K, Ali Darendeliler M, Swain M, Li Q. Computational and clinical investigation on the role of mechanical vibration on orthodontic tooth movement. J Biomech. 2017 Jul 26;60:57-64. doi: 10.1016/j.jbiomech.2017.06.012. Epub 2017 Jun 21. PMID 28743370